CLINICAL TRIAL: NCT03147664
Title: Cardiopulmonary Exercise Test to Quantify Enzyme Replacement Response in Pediatric Pompe Disease
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 3190-RMB-CTIL
Record Dates: First submitted 2017-04-30; First posted 2017-05-10 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Enzyme Replacement Therapy in Pompe Disease
Keywords: pompe disease; exercise capacity; cardiopulmonary exercise testing
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Pompe patients: Visit 1: Patients arrived at that hospital at 7:00 am, vital signs were collected and a complete neuromuscular evaluation was carried out (gross motor function measure score sheet (GMFM-88), 6MWT, pre-CPET questionnaire (demographics, physical activity level, risk assessment, asthma/atopy/smoking history, family history), pulmonary function tests and CPET. Following the evaluation, at approximately 9 am, the patient started infusion of ERT.
  Visit 2: Two days following visit 1, the patient arrived at the hospital at 2:00 pm, vital signs were assessed and GMFM-88, 6MWT, pulmonary function tests, and CPET were performed.

SUMMARY:
Introduction: Enzyme replacement therapy (ERT) with Myozyme improved the prospect of Pompe disease patients. Our aim was to evaluate ERT acute effect on exercise capacity in pediatric Pompe patients.

Methods: Pompe patients (10-19 years) were evaluated before and two days after ERT using cardiopulmonary exercise testing (CPET), six minutes walking test (6MWT) and motor function test (GMFM-88).

DETAILED DESCRIPTION:
Pompe disease is an inherited autosomal recessive glycogen storage disease caused by partial or total deficiency of acid α-glucosidase (GAA), resulting in the accumulation of glycogen in the lysosomes of skeletal muscles, heart, liver and other tissues. There is an inverse correlation between the amount of residual GAA activity and disease severity. The clinical phenotype varies with regard to age of onset, organ involvement, and severity of progression. In 2006, enzyme replacement therapy (ERT) with recombinant human GAA (Genzyme Corporation, Cambridge MA, USA) was approved and, since then, decisive modification of the course of the disease has been reported. Clinical studies in infants showed that ERT led to improvement in cardiac, respiratory and skeletal muscle functions, with achievement of independent walking, higher levels of physical activity, and survival beyond infancy.

Exercise capacity significantly affects Pompe patients' clinical picture and quality of life [5]. However, data on the effects of ERT on physiological variables related to exercise capacity is scarce. Cardiopulmonary exercise testing (CPET) is a well-known procedure to assess exercise capacity in adults and children in healthy and chronic conditions. Little is known regarding exercise capacity in the pediatric Pompe population. Our aim was to evaluate the acute effect of ERT on exercise capacity and different physiological variables in pediatric Pompe patients.

Patients were evaluated before and two days after ERT (20mg/kg/EOW). Each evaluation included CPET, pulmonary function tests, 6MWT and GMFM-88. All tests were carried out by the same experienced physician, exercise physiologist, and physiotherapist.

Visit 1: Patients arrived at that hospital at 7:00 am, vital signs were collected and a complete neuromuscular evaluation was carried out (gross motor function measure score sheet (GMFM-88), 6MWT, pre-CPET questionnaire (demographics, physical activity level, risk assessment, asthma/atopy/smoking history, family history), pulmonary function tests and CPET. Following the evaluation, at approximately 9 am, the patient started infusion of ERT.

Visit 2: Two days following visit 1, the patient arrived at the hospital at 2:00 pm, vital signs were assessed and GMFM-88, 6MWT, pulmonary function tests, and CPET were performed.

ELIGIBILITY:
Inclusion Criteria:

* Pompe disease diagnosed by a deficiency of acid alpha-glucosidase enzyme activity in dry blood spot and/or lymphocytes, followed by the study of the disease-causing mutations using DNA analysis of the GAA gene
* Age ≥8 y/o
* ERT ≥1 year
* Capable of cycling on a stationary bicycle.

Exclusion Criteria:

* Invasive ventilation
* Continuous ventilation and/or continuous oxygen supplementation to maintain oxygen saturation >90%
* Acute illness on visit day or one day prior.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric Pompe patients diagnosed by a deficiency of acid alpha-glucosidase enzyme activity in dry blood spot and/or lymphocytes, followed by the study of the disease-causing mutations using DNA analysis of the GAA gene. Age ≥8 y/o, ERT ≥1 year, capable of cycling on a stationary bicycle.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change in oxygen Uptake | 3 days
  Change in mount of oxygen consumed per amount of time measured during 15 minutes of an exercise test.

SECONDARY OUTCOMES:
6 Minute walk test | 3 days
  The distance an individual walked in 6 minutes.
Gross motor function measure score sheet (GMFM-88) | 3 days
  The patient is evaluated in the active performance of 88 physical tasks and the scoring range for each task ranges from 0=does not initiate, 1=initiates, 2=partially completes, 3=completes, NT=not tested. The total score is the sum of all tasks divided to the maximal potential score in percentage. Evaluation time ~ 30 minutes.
Spirometry | 3 days.
  Pulmonary function as assessed by spirometry. Evaluation time - 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No